CLINICAL TRIAL: NCT02186379
Title: Eating Pace Retraining in Childhood Obesity Prevention
Brief Title: Eating RePace Study
Acronym: REPACE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 12-009540
Record Dates: First submitted 2014-07-08; First posted 2014-07-10 (Estimated); Last update posted 2015-04-24 (Estimated); Status verified 2015-04

CONDITIONS: Obesity; Rapid Eating Style
Keywords: Obesity; Obesity Prevention; Childhood obesity prevention; Rapid Eating Style
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- RePace Intervention Group (Experimental): Re-Pace intervention-five weekly intervention sessions lasting about 1 hour each.
  Lab Test Meal-2 test meals 6-8 weeks apart.
  Interventions: Behavioral: RePace Intervention
- Usual Care Control Group (Active Comparator): One 25 minute education session (week 6) 2 lab test meals 6-8 weeks apart (baseline and week 6)
  Interventions: Behavioral: Usual Care Control

INTERVENTIONS:
Behavioral: RePace Intervention — The Re-Pace intervention will provide children and parents/caregivers training in strategies to promote slower eating pace and greater awareness of satiety levels. These skill building strategies can be classified as follows: 1) learning to slow eating rate, 2) awareness-raising activities; 3) role play activities; 4) self-monitoring training; 5) goal setting challenges; and 6) parent training. A core strategy for achieving slower eating pace and improved satiety will be to increase fruit and vegetable intake to meet United States Department of Agriculture (USDA) guidelines (www.myplate.gov). There are 5 intervention visits lasting about 1 to 1.25 hours each. See Section 4.3.1 for more details of the Re-Pace intervention.
  Arms: RePace Intervention Group
Behavioral: Usual Care Control — Following the second test meal session, parents and children will receive a brief (25 minute) instruction on healthy eating using materials from www.ChooseMyPlate.gov site, including "What's on Your Plate" and "My Plate for Kids" mini-posters.
  Arms: Usual Care Control Group

SUMMARY:
The aims of this study are to develop a novel family-based behavioral intervention (Re-Pace) to help children at risk for obesity (children who eat rapidly and have an overweight parent/legal guardian) develop a more normal eating rate.

DETAILED DESCRIPTION:
Childhood obesity is one of nation's foremost public health epidemics, for which more potent and enduring prevention interventions are needed. The goal of this program of research is to study novel methods which may help to prevent childhood obesity. The purpose of this randomized, controlled pilot study is to retrain children at risk for obesity (4-7 years of age in the 65th - <96th BMI percentile for age and sex, who have rapid eating and an obese participating parent/legal guardian [ N = 15]) to reduce their rate of eating (mouthfuls/minute) during a laboratory test meal, compared with participants in usual care control condition (UCC),which receives a brief educational intervention to promote healthy eating after the final assessment) (N=15). Between group change scores in mouthfuls/min (baseline Lab meal 1 to Lab meal 2) will be assessed. The investigators hypothesize that the children in the Re-Pace group will have a greater reduction in the rate of eating (mouthfuls of food/min) from baseline to week 6, compared to those in the UCC group.

As the sample size is relatively small, the aim is to develop an "effect size estimation," i.e., to generate an effect size that will be used to power an extramural grant application. Specifically, the investigators will generate Cohen's D as the effect size estimate, which is calculated as the difference in the group means divided by the pooled standard deviation. Cohen's D is an established quantitative measure for effect size estimation and informing power analysis for study design.

In addition, this study's objective is to develop and pilot a novel family-based eating behavior program for a prevention intervention in at risk children.

ELIGIBILITY:
Inclusion Criteria:

Children:

* Males or females 4 to 7 years of age.
* Participants (the children) have a body mass index (BMI) for age and sex between the 65th-<96th percentile (thus, the children will not have a BMI at the 97th percentile or more).
* Parental/guardian permission (informed consent).
* Have an overweight or obese participating parent/guardian with a BMI of > 27 kg/m2
* Increased child eating rate as reported on the questionnaire (Child Eating Behavior Questionnaire) by the parent/guardian

Parents:

* Parent/legal guardian of subject.
* Age 21 years and above.
* Have a BMI of > 27 kg/m2.

Exclusion Criteria:

Children:

* Children who have any developmental, medical, or psychiatric condition which might affect study compliance, as described by parental (caregiver) report.
* Children who have serious medical conditions or use of medications (e.g., chronic oral steroids, antipsychotic medications) known to affect food intake or body weight, as described by parental report.
* Children who have food allergies which may influence consumption of test foods, as reported by the parent; any child with reported peanut allergy.
* Parents/guardians or subjects who, in the opinion of the Investigator, may be non-compliant with study schedules or procedures.

Parents:

* Parents/guardians who, in the opinion of the Investigator, may be non-compliant with study schedules or procedures.

Ages: 4 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 28 (Actual)
Dates: Start 2012-11; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Reduction of eating rate (mouthfuls/min) | 6 weeks
  The purpose of this randomized, controlled pilot study is to retrain children at risk for obesity (4-7 years of age in the 65th - <96th BMI percentile for age and sex, who have rapid eating and an obese participating parent/legal guardian [ N = 15]) to reduce their rate of eating (mouthfuls/minute) during a laboratory test meal, compared with participants in usual care control condition (UCC),which receives a brief educational intervention to promote healthy eating after the final assessment) (N=15). Between group change scores in mouthfuls/min (baseline Lab meal 1 to Lab meal 2) will be assessed. We hypothesize that the children in the Re-Pace group will have a greater reduction in the rate of eating (mouthfuls of food/min) from baseline to week 6, compared to those in the UCC group.

SECONDARY OUTCOMES:
Reduction of food consumption | 6 weeks
  Reduce the rate of food consumption (kcal/min) and total kcal intake during the test meals (baseline Lab Meal 1 to Lab Meal 2). We also aim for participants to consume more fruits and vegetables during the test meal (baseline to week 6).

CONTACTS AND LOCATIONS:
Overall Officials: Robert I Berkowitz, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Faith MS, Diewald LK, Crabbe S, Burgess B, Berkowitz RI. Reduced Eating Pace (RePace) Behavioral Intervention for Children Prone to or with Obesity: Does the Turtle Win the Race? Obesity (Silver Spring). 2019 Jan;27(1):121-129. doi: 10.1002/oby.22329. Epub 2018 Dec 4. PMID 30515992